CLINICAL TRIAL: NCT05319210
Title: Investigation of the Effect of Virtual Reality Glasses and Buzzy Application on Pain Management During Venous Catheter Insertion in Children
Brief Title: The Effect of Virtual Reality and Buzzy Application on Pain Management in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Serife Tutar, Principal investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 188972
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Pain Management
Keywords: pain; virtual reality glasses; buzzy application; children; venous catheter
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy application (Experimental): It is fixed on the right upper arm area of the child one minute before the procedure. After cleaning the skin with the appropriate solution, venous catheter placement will be performed. During the procedure, the child's respiratory rate, heart rate and oxygen saturation will be observed.
  Interventions: Procedure: Venous catheter application
- Virtual Reality Glasses (Experimental): A dinosaur movie suitable for the 7-12 age group will be watched 2-3 minutes before the venous catheter insertion. In this process, after cleaning the skin with the appropriate solution, a venous catheter will be inserted. During the procedure, the child's respiratory rate, heart rate and oxygen saturation will be observed.
  Interventions: Procedure: Venous catheter application
- No intervention (No Intervention): The routine venous catheter placement protocol in the institution where the study is conducted will be applied. An evidence-based non-pharmacological method is not used to reduce pain during venous catheter insertion in children in the institution. A venous catheter is inserted by attaching a tourniquet to the child. During the procedure, the child's respiratory rate, heart rate and oxygen saturation will be observed.

INTERVENTIONS:
Procedure: Venous catheter application — To examine the effect of virtual reality glasses and buzzy application on pain management during venous catheter insertion in children.
  Arms: Buzzy application; Virtual Reality Glasses

SUMMARY:
The purpose of this research; This is a randomized controlled experimental study planned to examine the effect of virtual reality glasses and buzzy application on pain management during venous catheter insertion in children.

DETAILED DESCRIPTION:
The purpose of this research; This is a randomized controlled experimental study planned to examine the effect of virtual reality glasses and buzzy application on pain management during venous catheter insertion in children.

The universe of the research is all children between the ages of 7 and 12 who applied to Hospital Emergency Service will be formed. G power analysis program was used to calculate the sample size of the study. The number of samples was calculated according to 95% power, 0.05 margin of error and 0.80 effect size. It is envisaged that 36 children will be included in the sample for each group. However, considering that sample losses may be experienced during the process of the research, it is planned to include 40 participants (120 participants in total) for each group.

"Child and Parent Diagnosis Form", "Child Fear Scale (CDS)", "Child Anxiety Scale-State (CAS-D)" and Wong-Baker Faces Pain Scale will be used to collect research data.

In the collection of research data, first of all, patients will be divided into intervention and control groups in accordance with the randomization scheme. Our research will consist of two interventions (Buzzy device, virtual reality glasses) and a control group (routine outpatient procedures).

Before the procedure; Written and verbal "Informed Consent" will be obtained from all participants in the intervention and control groups. "Child and Parent Diagnosis Form", "Child Fear Scale (CDS)", "Child Anxiety Scale-State (CAS-D)" and Wong-Baker Faces Pain Scale will be applied to the participants who agree to participate in the study.

Process Sequence and After; Venous catheter insertion will be done in line with the routine practice of the outpatient clinic. Venous catheter placement in all children included in the study will be performed by the researcher working in this one in order to keep the practitioner-related factors under control. Children who cannot insert a venous catheter in a single attempt will be excluded from the study.

Licensed SPSS (Statistical Package for the Social Science) 20.0 package program will be used in the evaluation of the data. Descriptive analyzes such as number, percentage, frequency, mean, standard deviation and percentile distributions will be used to evaluate the characteristics of children. Nonparametric tests will be used according to the results of normal distribution and homogeneity of variance. Mann Whitney U test, Wilcoxon test and correlation analyzes will be used to evaluate the relationships between dependent and independent variables. Results will be evaluated at 95% confidence interval and p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the research
* 7-12 age group
* The child does not have vision, hearing, mental or neurological sequelae.

Exclusion Criteria:

-Children with a history of using sedative, analgesic or narcotic substances with analgesic effect before admission to the outpatient clinic will not be included in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain management | 4 month
  Management of pain during venous catheter insertion in children. The parameter for pain management will be determined by the Wong Baker Faces Pain Rating Scale.

SECONDARY OUTCOMES:
Management of fear in children | 4 month
  Management of fear during venous catheter insertion in children. The parameter for fear management will be determined by the Child Fear Scale.
Management of anxiety in children | 4 month
  It is the management of anxiety during venous catheter placement in children. The parameter for Anxiety management will be determined by Child Anxiety Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Tutar T Assistant professor, PhD, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No